CLINICAL TRIAL: NCT05992285
Title: A Randomized, Controlled Clinical Study of Continuous Theta Burst Stimulation (cTBS) in the Treatment of Insomnia Disorder Targeting the Dentate Nucleus of the Cerebellum
Brief Title: A Clinical Study of Theta Burst Stimulation (cTBS) in the Treatment of Insomnia Disorder Targeting the Dentate Nucleus of the Cerebellum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20232190
Record Dates: First submitted 2023-07-17; First posted 2023-08-15 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cTBS group (Experimental): the intensity of stimulus was 80% Resting motor threshold (RMT); the frequency of trains was 50 Hz and the number of pulses was three; and the frequency of intertrain intervals was 5 Hz and pulses number was 200. Two groups were repeatedly stimulated in the dentate nucleus of bilateral cerebellum, the interval of each group was 5min, and the number of stimulation pulses at each site was 1200.
  Interventions: Device: transcranial magnetic stimulation
- sham group (Sham Comparator): The treatment of the sham group was the same as active group. The only difference was that the coil was flipped 180° in the sham group. The device also made the same sound but could not stimulate the brain.
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — the intensity of stimulus was 80% Resting motor threshold(RMT); the frequency of trains was 50 Hz and the number of pulses was three; and the frequency of intertrain intervals was 5 Hz and pulses number was 200. Two groups were repeatedly stimulated in the dentate nucleus of bilateral cerebellum, the interval of each group was 5min, and the number of stimulation pulses at each site was 1200.

SUMMARY:
Insomnia disorder (ID) is a significant public health problem worldwide, with nearly a third of the general population experiencing insomnia symptoms in their lifetime. Therefore, finding a safe, effective, and easy-to-use non-pharmacological method for treating ID is urgent. Repetitive transcranial magnetic stimulation (rTMS) has been used to varying degrees in many neurological and psychiatric diseases and has broad application prospects for treating ID.θ-burst stimulation is characterized by cluster stimulation.Continuous stimulation (cTBS) mainly has inhibitory effects on the cortex. The inhibition of motor-evoked potentials can last for 60 minutes, which is longer-lasting, has a lower stimulation intensity, and is shorter in duration than traditional rTMS. There are no reports on clinical studies of cTBS treatment for ID. So far, sleep research has mainly focused on the interconnections between the neocortex and subcortical structures, while cerebellar activity has been largely overlooked.The mechanism of rTMS treatment for insomnia with the cerebellum as the target is unclear. This study proposes to apply cTBS mode to the cerebellar dentate nucleus for rTMS treatment in patients with ID to explore its effectiveness and safety in improving insomnia disorder.

ELIGIBILITY:
Inclusion Criteria:

* All participants aged from 18 to 60 years old; all participants met diagnostic criteria for insomnia disorder according to the Diagnostic and Statistical Manual of Mental Disorders-V (DSM-V), and scored >10 on PSQI , ≤14 on the Hamilton Anxiety Scale (HAMA), and ≤17 on the Hamilton Depression Scale (HAMD); no sleep-affecting drugs were taken 1 month before or during the trial (non-prescription sleep medication, benzodiazepines or hypnotics, ect.); patients can cooperate to complete the treatment and related examination items; all subjects signed informed-consent forms before enrolling in the trial.

Exclusion Criteria:

* The patient is unable to cooperate with the completion of treatment and examinations; there are other types of sleep disorders; a history of psychotropic drug or alcohol dependence or abuse in the last 2 years; have undertaken trans-meridian travel across more than two time zones or worked night shifts in the preceding one month or during the trial period; plan surgical treatment within 1 month before or during the trial; evidence of neurological or other physical diseases such as respiratory, cardiac, renal, hepatic, endocrinal diseases and other psychiatric diseases as assessed by clinical history, physical examination or routine laboratory tests; pregnancy or breastfeeding women; any contraindication for rTMS (including implanted metal and devices in the body, and history of epilepsy); concurrent other clinical trials; patient or family member withdraws informed-consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
The reduction rate of the Pittsburgh Sleep Quality Index（PSQI） score | At the end of 10 days of treatment
  The reduction rate of the Pittsburgh Sleep Quality Index (PSQI) score

SECONDARY OUTCOMES:
Improvement rate of polysomnography monitoring index | At the end of 10 days of treatment and 1 month follow-up
  Improvement rate of polysomnography monitoring index, including total sleep time, fall asleep time, wake time, sleep efficiency, sleep structure, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Air Force Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No